CLINICAL TRIAL: NCT03151460
Title: Dopaminergic Modulation of Declarative Memory
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Giovanni Augusto Carlesimo, Professor, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Dopamine Agents

STUDY DESIGN:
Intervention Model Description: All PD patients were examined in two conditions: following the standard dopamineric medication ("on") and following a 12-18 hours of treatment wash-out ("off"). Normal controls were examined twice with no drug assumption.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson (Experimental): Patients with Parkinson's disease assuming or not Dopamine Agents
  Interventions: Drug: Dopamine Agent
- Normal Controls (No Intervention): Age and education comparable healthy subjects

INTERVENTIONS:
Drug: Dopamine Agent — Patients were assessed in two experimental conditions that were performed on different days, with an intersession interval of about one month. In the "off" condition PD subjects performed the experimental tasks in the morning after 12/18 hours of Dopamine Agent withdrawal. In the "on" condition they were examined 90-120 minutes after they had taken their first morning dose of levodopa and/or dopamine agonists.
  Other Names: Dopaminergic drugs
  Arms: Parkinson

SUMMARY:
The study investigates the effect of dopaminergic stimulation over declarative memory functions in Parkinson's disease (PD) patients. At this aim, 20 PD patients will receive declarative memory tasks in two different conditions: after 12-18 hours of dopaminergic stimulation withdrawal ("off" condition) and after the first daily dose dopaminergic therapy ("on" condition). 20 healthy controls will also administered the two tasks in two conditions with the same inter-session delay as PD patients, but without taking drugs.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is frequently accompanied by declarative memory deficits. It has been hypothesized that these latter could be related to dopaminergic depletion within the fronto-striatal network. However, the nature of this relationship is not clearly understood. In this study we aim to assess the role of daily dopaminergic stimulation on the retrieval processes needed to perform different cognitive tasks. A group of PD patients will be administered declarative memory task both "on" (standard medication intake) and "off" (12/18 hours after the last medication intake). A group of comparable normal controls will also present with the same cognitive task twice, without any drug assumption. Understanding the effect of dopamine treatment on declarative memory processes will allow standard medication treatment to be adjusted in order to take into account both motor and cognitive features of Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson Disease made by a neurologist according to the London Brain Bank criteria.

Exclusion Criteria:

* disease duration ≥ 5 years; diagnosis of dementia based on clinical criteria and confirmed by a Mini-Mental State Examination score < 26; presence of other neurological and/or psychiatric illnesses in the patient's clinical history.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Performance on cognitive task | 60 min.
  Performance scores on declarative memory tasks

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Carlesimo, MD, Principal Investigator — Fondazione S. Lucia
Locations (1):
- Fondazione S. Lucia, Rome, Italy

IPD SHARING:
Plan to Share IPD: No